CLINICAL TRIAL: NCT05142384
Title: ICBT for Maternal Depression: Community Implementation in Head Start
Brief Title: ICBT (Internet Based Cognitive Behavioral Therapy) for Maternal Depression: Community Implementation in Head Start
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH120237
Record Dates: First submitted 2021-09-29; First posted 2021-12-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics; Waiting Lists

STUDY DESIGN:
Intervention Model Description: Head Start (HS) agencies will be randomized to offer Mom-Net with either high- or low- intensity coaching. Subsequently, participants will be randomized to either the Mom-Net condition offered by their child's HS agency or to Treatment as Usual within the community/Waitlist (TAU/WL). Assessments will be conducted at T1- prior to participant randomization, at T2- subsequent to the conclusion of the intervention period, and at T3 1 year after T1. Subsequent to the T2 assessments, participants in the TAU/WL condition will be offered the opportunity to participate in the Mom-Net version offered by their HS agency. The T3 assessment will thus enable us to examine Maintenance of effects for those in the Mom-Net condition, and Replication of Mom-Net within group effects for those in the TAU/WL condition.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to participant condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mom-Net (Experimental): Mom-Net is a guided Internet intervention. Mom-Net is distinct from other CBT interventions for depression in addressing the link between maternal depression and parenting. Mom-Net's content includes core CBT skills taught in ways that are relevant to one's parenting interactions. Mothers will participate in Mom-Net with either high- or low-intensity coaching as determined by which version their HS was randomized to offer. Coaching is provided by HS staff.
  In the high-intensity version, coaches provide support both for engaging with the intervention and for learning content. Coaching phone calls occur weekly (20-30 min call per session). In the low-intensity version, coaches provides supportive accountability for engaging with the intervention. Mothers participate in 4 (10-15) min calls occurring post-randomization, and 3- and 6-weeks later.
  Interventions: Behavioral: Mom-Net
- Treatment as Usual/Waitlist (Active Comparator): HS sites provide ongoing social and instrumental support to parents, including helping to connect families to needed services including community mental health providers. Additionally, research staff will provide lists of local mental health providers and information to support treatment seeking. Research staff will also provide National Crisis Lines for Mental Health Emergencies. Staff will inform participants to call research staff if they have trouble accessing services so that staff may provide additional help. Finally, staff will share a case note documenting referrals with the women's family service worker, so that worker may provide locally based assistance to the woman in accessing services. Subsequent to T2 assessment, participants in the TAU/Waitlist condition, will be offered the Mom-Net intervention variant (high- v low-intensity coaching) being provided by their respective HS agencies.
  Interventions: Combination Product: Treatment as Usual/Waitlist

INTERVENTIONS:
Behavioral: Mom-Net — Mom-Net is a guided Internet intervention. Mom-Net is distinct from other CBT interventions for depression in addressing the link between maternal depression and parenting. Mom-Net's content includes core CBT skills taught in ways that are relevant to one's parenting interactions. Mothers will participate in Mom-Net with either high- or low-intensity coaching as determined by which version their HS was randomized to offer. Coaching is provided by HS staff.
  In the high-intensity version, coaches provide support both for engaging with the intervention and for learning content. Coaching phone calls occur weekly (20-30 min call per session). In the low-intensity version, coaches provides supportive accountability for engaging with the intervention. Mothers participate in 4 (10-15) min calls occurring post-randomization, and 3- and 6-weeks later.
  Arms: Mom-Net
Combination Product: Treatment as Usual/Waitlist — HS sites provide ongoing social and instrumental support to parents, including helping to connect families to needed services including community mental health providers. Additionally, research staff will provide lists of local mental health providers and information to support treatment seeking. Research staff will also provide National Crisis Lines for Mental Health Emergencies. Staff will inform participants to call research staff if they have trouble accessing services so that staff may provide additional help. Finally, staff will share a case note documenting referrals with the women's family service worker, so that worker may provide locally based assistance to the woman in accessing services. Subsequent to T2 assessment, participants in the TAU/Waitlist condition, will be offered the Mom-Net intervention variant (high- v low-intensity coaching) being provided by their respective HS agencies
  Arms: Treatment as Usual/Waitlist

SUMMARY:
Low income women of childbearing age are at increased risk for depression and often do not receive needed treatment. Investigators developed Mom-Net, an on-line cognitive behavioral treatment (CBT) for depression to address the needs of low income women of childbearing age. The intervention program also includes live coaching to help the mothers engage and learn the CBT material. Mom-Net has been shown to be highly effective in reducing depressive symptoms and improving parenting behavior and child adjustment, in earlier controlled trials. In this project the investigators are examining whether access to Mom-Net can be expanded by delivering it in Head Starts (HS).

To address that broad question, the investigators will focus on two sets of scientific questions:

1. Implementation Questions: e.g., Can HS agencies deliver the program successfully; do HSs choose to sustain the program after the research project ends; what agency characteristics are associated with successful delivery of Mom-Net);
2. Effectiveness Questions: e.g., Does Mom-Net reduce maternal depression when delivered by Head Start agencies, with HS staff doing the coaching?

Head Start agencies will be randomized to deliver either Mom-Net with the usual high-intensity coaching or with a low-intensity coaching alternative. Within each agency, depressed mothers will be randomized to receive either: 1) Mom-Net program; or 2) Treatment as Usual (TAU;) referral to community mental health providers). Mothers initially assigned to the TAU condition, will have the option of receiving Mom-Net at a later date. Mothers will participate in assessments of depressive symptoms, parenting behavior, and child adjustment at Time 1 (T1; prior to randomization); and Time 2 (T2; after the intervention period) and Time 3 (T3; one year after T1).

DETAILED DESCRIPTION:
Background:

Low income women of childbearing age are at disproportionate risk for depressive syndromes and, despite the availability of efficacious interventions, often do not receive needed treatment. The investigators developed Mom-Net, a remote, coach-facilitated, Internet-based intervention adapted from an empirically-supported cognitive behavioral treatment (CBT) for depression to address the needs of depressed mothers. Two randomized control trials demonstrated Mom-Net to be highly effective in reducing depressive symptoms and improving parenting behavior and child adjustment. In this project investigators seek to examine whether the reach of the Mom-Net intervention can be expanded by implementing within the Head Start Environment.

Investigators are using a hybrid type 2, Effectiveness-Implementation design to compare two implementation approaches for the delivery of Mom-Net, one with its existing high-intensity coaching approach, and one making use of a low-intensity coaching, designed to provide supportive accountability, but not psychoeducational support. Investigators will follow the Exploration, Preparation, Implementation, and Sustainment process model (EPIS) to guide the evaluation, with the Clinical Trial component primarily constituting the Implementation phase.

Clinical Trial Aims:

1. Examine effectiveness and Implementation outcomes of Mom-Net within Head-Start, randomizing agencies to implementation approach (i.e., high- vs low-intensity coaching) and mothers within agency, to either Mom-Net or Treatment as Usual (TAU)/waitlist conditions.

   1. Compare the two Mom-Net implementation approaches on: 1) implementation outcomes including reach, acceptability, fidelity, and cost; and 2) effectiveness outcomes including self-reported maternal depressive symptoms (primary outcome), parenting behavior, and child emotional and behavioral functioning (secondary outcomes).
   2. Examine the effectiveness of each Mom-Net implementation approach relative to TAU on the primary and secondary outcomes listed above.
2. Consistent with an experimental therapeutic approach, investigators will examine the mediating influence of changes in maternal functioning associated with core Mom-Net skills on maternal depressive symptoms. Mediators to be examined include behavior activation, negative cognitive styles, social support, and belief that mood can be regulated. Investigators will also examine the mediating influence of change in maternal depressive symptoms on parenting behavior and child outcomes.

Clinical Trial Protocol

1. Prior to the Implementation Phase (i.e., clinical trial), participating agencies will be randomized to either high- or low-intensity coaching conditions.

ELIGIBILITY:
Inclusion Criteria: Mothers

* Elevated symptoms of depression (i.e., Patient Health Questionnaire or Edinburgh Postnatal Depression Scale score at or above 10)
* Have a child 2-5 years enrolled in a participating Head Start; be able to communicate in English or Spanish.

Inclusion Criteria: Child

- 2-5 years of age and enrolled in participation Head Start

Exclusion Criteria: Mothers

* Evidence of psychosis or other major mental illness or cognitive disability (observed during recruitment or by HS report) that would interfere with meaningful participation
* Endorsed score of 3 on final item of the PHQ9 or EPDS indicating frequent thoughts of suicide. Could be enrolled at later date if elevated risk ameliorates

Exclusion Criteria: Children

* No exclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Assessing change between baseline, post-intervention (5 months), and follow up (12 months)
  Well-established measure of maternal depression with 9 self-report items, each rated on a 0 (not at all) to 3 (nearly every day) scale; total score will be used; interpretation: scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe,and severe depression, respectively. Total score will be used to examine change from baseline to subsequent assessments.
Maternal Acceptability (Modified System Usability Scale) | Post intervention ( 5 months)
  Implementation Outcome Variable. 14-item scale, rated on a 1-5 response scale. Will examine perceived helpfulness of Mom-Net content, activities, and coach calls. This scale has been used in investigators' prior Mom-Net research. The summed-item total score will be used, with a scale range of 14-70.
Screening Reach (Reach) | End of screening in year 2 of implementation
  Implementation Outcome. Screening rates will be calculated as the number of PHQ-9 screeners administered within each agency each year divided by the family HS enrollment (with a female-identified parent-figure). The metric will represent the percentage of mothers in each agency who were reached, with a range of 0-100.
Implementation Reach (IReach) | End of Implementation in Year 2
  Implementation Outcome. Calculated as the number of Mom-Net eligible mothers screened within each agency divided by the number of mothers within each agency initiating Mom-Net intervention with a within-agency range of 0-100%.
Maternal Engagement (Engage) | Change between base-line and 5-month assessments
  Number of modules (0-8) and coach calls completed, page views (0-120), and program visits (0- no upper limit). These well-established indices of usage will be collected in real time.

SECONDARY OUTCOMES:
Parent Behavior Inventory (PBI) | Change between Baseline and 5- and 12-month follow-up
  Subscales will all be used to examine change in maternal behavior from baseline through subsequent assessment points; subscale total scores will be used; all items rated on a 0 (I don't do this) to 5 (I often do this) scale and summed for subscale total; Supportive/Engaged sub-scale range 0-55, Hostile/Coercive subscale range 0-45.
Parenting Sense of Competence (PSOC) | Change between Baseline and 5- and 12-month follow-up
  Will use will three metrics to assess change in maternal sense of competence from Baseline through subsequent assessments: Total score, 17 items; Efficacy subscale, 8 items, Valuing/Comfort subscale, 9 items; all items are rated on a 1 (Strongly Agree) to 6 (Strongly Disagree) scale. Items will be summed to form: Total score (range of 17-102), Efficacy score (range 4-48) and Valuing/Comfort score (range 9-54). For total and subscale scores, a high score will reflect strong competence.
Child Behavior Checklist (CBCL 1 ½ - 5 years) | Change between Baseline and 5- and 12-month follow-up
  Well-established measure of child internalizing/externalizing behavior; all items rated on 0 (not true), 1 (somewhat or sometimes true), 2 (very true or often true) scale; Both the Internalizing (36 items) and externalizing (24 items) subscales will be used, with raw score ranges of 0-72 and 0-48, respectively. Raw scores will be used in analysis of the age-associated t-scores.
Child Behavior Checklist Teacher Report Form (C-TRF) | Change between Baseline and 5- and 12-month follow-up
  Well-established measure used to examine change in child internalizing/externalizing behavior; all items rated on 0 (not true), 1(somewhat or sometimes true), 2 (very true or often true) scale; Both the internalizing (32 items) and externalizing (34 items) subscales will be used, with raw score ranges of 0-64 and 0-68, respectively. Will be used in analysis of the t-scores associated with the raw score totals.
Aggressive Interpersonal Behavior (Proportion) | Change between Baseline and 2-4 month assessment
  The Living in Family Environments (LIFE) and Dyadic Parent-Child Interaction Coding System (DPICS) are two systems for coding family interactions. Investigators are using the LIFE affective codes and the DPICS verbal codes. Though the LIFE has verbal codes, the DPICS verbal codes are more developmentally appropriate. This approach has been used in earlier work. This outcome reflects the proportion of aggressive interpersonal behavior across the duration of the interaction.
Aggressive Interpersonal Behavior (Duration) | Change between Baseline and 2-4 month assessment
  The Living in Family Environments (LIFE) and Dyadic Parent-Child Interaction Coding System (DPICS) are two systems for coding family interactions. Investigators are using the LIFE affective codes and the DPICS verbal codes. Though the LIFE has verbal codes, the DPICS verbal codes are more developmentally appropriate. This approach has been used in earlier work. This outcome reflects the duration per episode of aggressive interpersonal behavior observed during the interaction.
Positive Interpersonal Behavior (Proportion) | Change between Baseline and 2-4 month assessment
  The Living in Family Environments (LIFE) and Dyadic Parent-Child Interaction Coding System (DPICS) are two systems for coding family interactions. Investigators are using the LIFE affective codes and the DPICS verbal codes. Though the LIFE has verbal codes, the DPICS verbal codes are more developmentally appropriate. This approach has been used in earlier work. This outcome reflects the proportion of positive interpersonal behavior across the duration of the interaction.
Positive Interpersonal Behavior (Duration) | Change between Baseline and 2-4 month assessment
  The Living in Family Environments (LIFE) and Dyadic Parent-Child Interaction Coding System (DPICS) are two systems for coding family interactions. Investigators are using the LIFE affective codes and the DPICS verbal codes. Though the LIFE has verbal codes, the DPICS verbal codes are more developmentally appropriate. This approach has been used in earlier work. This outcome reflects the duration per episode of positive interpersonal behavior observed during the interaction.
The Work and Social Adjustment Scale | Change between Baseline and 2-4 month assessment
  The Work and Social Adjustment Scale (WSAS) assesses the impact of mental health diﬃculties on ability to function in the context of work, home management, social leisure, private leisure, and personal or family relationships. Possible scores range from 0 to 40, where lower scores indicate fewer symptoms.
5-item World Health Organization Well-Being Index | Change between Baseline and 2-4 month assessment
  The Well-Being Index is a short self-report measure assessing current wellbeing. Possible scores range from 0 to 25, where higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Edward G Feil, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participant data will be available through the National Institute of Mental Health (NIMH) Data Archive (NDA)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be loaded into NDA every 6 months once recruitment begins.
Access Criteria: Compliant with NIMH NDA requirements